CLINICAL TRIAL: NCT00616369
Title: Identification of Genetic Markers for Cardiopulmonary Diseases
Brief Title: Identification of Genetic Markers for Cardiopulmonary Diseases (Genotype)
Acronym: Genotype
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: X070116004
Record Dates: First submitted 2008-02-05; First posted 2008-02-15 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Cardiovascular Diseases
Keywords: pulmonary hypertension; hypertension; cardiomyopathy; arrhythmias
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension, Pulmonary; Hypertension; Cardiomyopathies; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The following genetic tests will be performed on these specimens:
  Endothelin1, Endothelin receptors A&B, Prostaglandin, Prostaglandin receptors, CytochromeP450, NPR, A, B and C, Transforming Growth Factor (B), Pai-1 HindIII, Toll-like receptor4, Pai-1 4g5g, Xho-1, P22, Tissue Plasminogin Activators, Urokinase Plasminogen Activators, Fibrinogen, Nitric Oxide Synthase, BMPRs, SMADs, VEGFs, FGFs, Rho Kinase, Elastins, Angiopoietin, PDE5, Serotonin receptor, Angiotensin, Alk 1, and Cell Culture (DNA immortalization)
  There is a possibility that other genetic testing could arise as the study progresses. In this case, the IRB would be notified prior to testing.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: I:
  For those patients who have had blood samples drawn as a result of participating in current protocol, Identification of Genetic Markers for Primary Pulmonary Hypertension study (X980515002), we would like to use their previously obtained blood and continue to draw samples (12mL; less than 3 tablespoons) ONLY if they change disease therapies.
  For those patients who participated in Pulmonary Arterial Hypertension (PAH) Database study (X030403017), these participants will also sign a consent form to participant in this new trial. We would like to use the previously obtained data from the X030403017 in part with this study.
  As for the X980515002 expired patients, we would like to use the previously obtained data ONLY in part for this study that was collected as a result of the X980515002 study.
- 2: II:
  Group 2: After signing a consent form, these participants will have a 12mL (less than 3 teaspoons) blood sample drawn at baseline, at 3-4 month, at 6-8 month, at 12 month, and at 24 month visits. With each disease therapy change, the blood draws (12mL samples) will begin again at baseline and continue through the 3-4, 6-8, 12, and 24 month visits.

SUMMARY:
This study is designed to investigate whether an association exists between certain genes/protein levels and the development of various cardiopulmonary diseases. It is hoped that this project will provide valuable insight into the understanding of these diseases.

DETAILED DESCRIPTION:
There are two main groups of participants in this trial:

Group 1: Patients that are enrolled in either or both of previous studies: X980515002 study (Identification of Genetic Markers for Primary Pulmonary Hypertension) and or X030403017 study (Pulmonary Arterial Hypertension (PAH) Database)

Group 2: Participants with the diagnosis of any of the previously listed Cardiopulmonary Diseases who are ≥15 years of age

Group 1: For those patients who have had blood samples drawn as a result of participating in the current protocol, Identification of Genetic Markers for Primary Pulmonary Hypertension study (X980515002), we would like to use their previously obtained blood and continue to draw samples (12mL; less than 3 tablespoons) ONLY if they change disease therapies. With each disease therapy change, blood will be drawn at baseline, at 3-4 month, at 6-8 month, at 12 month, and at 24 month visits. These current X980515002 participants WILL sign a consent form to participate in this new trial. As for the X980515002 expired patients, we would like to use the previously obtained data ONLY in part for this study that was collected as a result of the X980515002 study.

For those patients who participated in Pulmonary Arterial Hypertension (PAH) Database study (X030403017), these participants WILL also sign a consent form to participant in this new trial. We would like to use the previously obtained data from the X030403017 in part with this study. With each disease therapy change, a 12mL (less than 3 teaspoons) blood sample will be drawn at baseline, at 3-4 month, at 6-8 month, at 12 month, and at 24 month visits. As for the X030403017 expired patients, we would like to use the previously obtained data in part for this study that was collected as a result of the X030403017 study.

Group 2: After signing a consent form, these participants will have a 12mL (less than 3 teaspoons) blood sample drawn at baseline, at 3-4 month, at 6-8 month, at 12 month, and at 24 month visits. With each disease therapy change, the blood draws (12mL samples) will begin again at baseline and continue through the 3-4, 6-8, 12, and 24 month visits.

ELIGIBILITY:
Inclusion Criteria:

* Participants with the diagnosis of any of the previously listed Cardiopulmonary Diseases who are ≥15 years of age will be approached and offered the opportunity to participate in this study.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with the diagnosis of any of the previously listed Cardiopulmonary Diseases who are ≥15 years of age will be approached and offered the opportunity to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2008-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Changes in NYHA WHO Functional Class,right and left heart catheterization measurements, echocardiograms, 6MWT, laboratory values, electrocardiograms, x-ray's, MRI's, CT Scans, Pulmonary Function Tests, and Ventilation Perfusion Scans will be assessed. | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Bourge, MD, Principal Investigator — University of Alabama at Birmingham Division of Medicine
Locations (1):
- University of Alabama @ Birmingham, Birmingham, Alabama, United States